CLINICAL TRIAL: NCT06027814
Title: Patient Navigator Plus Remote mHealth Adherence Support With Incentives to Improve Linkage and Retention Among Hospitalized Patients With Opioid and Methamphetamine Use Who Initiate Buprenorphine
Brief Title: MHealth Incentivized Adherence Plus Patient Navigation
Acronym: MIAPP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Judith I. Tsui, Professor, School of Medicine, General Internal Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00016329; 1R34DA057609-01 (NIH)
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Medication Adherence; Polysubstance Drug Use (Indiscriminate Drug Use); Methamphetamine-dependence
MeSH Terms: conditions — Opioid-Related Disorders; Medication Adherence | interventions — Patient Navigation; Telemedicine

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to treatment group. Group assignment will occur through computerized (REDCap) randomization procedures. The investigators will stratify randomization by whether the patient has buprenorphine treatment in the past year. Randomization lists will be prepared within each stratum using random block sizes of 4 to ensure balanced groups throughout the enrollment period. Participants will be informed of their assignment by research staff after completion of informed consent and the baseline survey.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment-as-usual (TAU) (No Intervention): TAU will be usual care that the Addiction Consult Service provides. It is comprised of a multidisciplinary team of professionals, including addiction medicine and addiction psychiatry physicians, nurses specializing in the treatment of OUD, substance use disorder counselors, peer recovery supports, and program coordinators.
- PN+mHealth (Experimental): The intervention is patient navigation and mHealth in addition to treatment-as-usual. The intervention consists of a patient navigator (PN) with the mHealth adherence application facilitating telehealth visits, two-way chats, video-DOT, and delivery of financial incentives via smartphone for adherence and linkage to outpatient treatment within 30 days. Participants will be asked to upload medication adherence videos once a day over the 30 days post discharge from the hospital. Patients will be instructed to continue to take their medication as prescribed in any circumstance where they are unable to upload the video for any reason.
  Interventions: Behavioral: Patient Navigation and mHealth (PN+mHealth)

INTERVENTIONS:
Behavioral: Patient Navigation and mHealth (PN+mHealth) — Intervention consists of patient navigation with the mHealth adherence application facilitating telehealth visits, two-way chats, video-DOT, and delivery of financial incentives via smartphone.
  Arms: PN+mHealth

SUMMARY:
Polysubstance use involving opioids and methamphetamine is emerging as a new public health crisis. Patients with opioids and methamphetamine use often experience serious medical complications requiring hospitalization, which provides an opportunity to offer addiction treatment. Yet linkage to outpatient treatment post-discharge is suboptimal and methamphetamine exacerbates outcomes. The investigators propose to pilot test "MHealth Incentivized Adherence Plus Patient Navigation" (MIAPP) to promote treatment linkage and retention for patients with opioid use disorder (OUD) and methamphetamine use who initiate buprenorphine in the hospital. The investigators Aim is to perform a two-arm, pilot randomized clinical trial (n=40) comparing MIAPP + treatment-as-usual (TAU) versus TAU alone on outpatient medication for opioid use disorder (MOUD) linkage within 30 days (primary) and 90-day retention on medications (secondary) among hospitalized patients with OUD and methamphetamine use.

ELIGIBILITY:
Inclusion Criteria:

* Adult greater than or equal to 18 years of age
* Admitted to Harborview Medical Center (HMC) on any inpatient service
* Initiated on buprenorphine for OUD while in the hospital or at the time of discharge and planning to continue outpatient
* Used methamphetamine within the past 30 days (any route of administration or frequency)
* Willing to be randomized to video-DOT
* Willing and able to use a smartphone (study can provide) and work with patient navigator
* Discharge setting does not preclude the use of video-DOT (i.e., nursing home, inpatient psychiatry, etc.)

Exclusion Criteria:

* Unable or unwilling to use smartphone (phones to be provided when needed)
* Cognitive impairment (acute or chronic) resulting in inability to provide informed consent
* Currently incarcerated and will discharge to jail or prison
* Plans to discontinue buprenorphine in the near future (<3 months)
* Lives far away such that cannot keep study visit at 30 days post-discharge
* Not English speaking
* Behavioral risk per discretion of research staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2026-09-22 (Estimated)

PRIMARY OUTCOMES:
Patient linkage to an outpatient program that provides medication for opioid use disorder | 30 days post-discharge from hospital
  Defined as documentation of an outpatient clinical encounter (either in-person or via telemedicine) where a medication for OUD (either buprenorphine, naltrexone, or methadone) was provided or prescribed.

SECONDARY OUTCOMES:
Retention on medication for opioid use disorder | 90 days post-discharge from hospital
  This will be measured as the number of days with medication coverage. (buprenorphine, naltrexone, or methadone).
Hospital readmission | 90 days post-discharge from hospital
  The number of hospital admissions will be extracted from statewide Medicaid claims data.
Emergency department visits | 90 days post-discharge from hospital
  The number of emergency department visits will be extracted from statewide Medicaid claims data.
Past 30-day opioid use | 30 days post-discharge
  The number of days using illicit opioids in the past 30 days per self-report as collected through the modified Addiction Severity Index.
Past 30-day methamphetamine use | 30 days post-discharge
  The number of days using methamphetamine in the past 30 days per self-report as collected through the modified Addiction Severity Index.

CONTACTS AND LOCATIONS:
Overall Officials: Judith I Tsui, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bhatraju EP, Kennedy DN, Gojic AJ, Iles-Shih M, Merrill JO, Samet JH, Hallgren KA, Tsui JI. mHealth Incentivized Adherence Plus Patient Navigation (MIAPP): protocol for a pilot randomized controlled trial to improve linkage and retention on buprenorphine for hospitalized patients with methamphetamine use and opioid use disorder. Addict Sci Clin Pract. 2025 Jan 29;20(1):6. doi: 10.1186/s13722-025-00538-1. PMID 39881397